CLINICAL TRIAL: NCT04966234
Title: Prospective Validation and Clinical Evaluation of a New Posaconazole Dosing Regimen for Children and Adolescents With Cystic Fibrosis and Aspergillus Infection
Brief Title: A New Posaconazole Dosing Regimen for Paediatric Patients With Cystic Fibrosis and Aspergillus Infection
Acronym: cASPerCF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: University of Exeter (Other); Radboud University Medical Center (Other); Consorzio per Valutazioni Biologiche e Farmacologiche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cASPerCF_2007_OPBG_2019; 2019-004511-31 (EudraCT Number)
Record Dates: First submitted 2021-03-19; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis; Aspergillosis
Keywords: Posaconazole; Progressive lung damage; Recurrent infection; Persistent inflammation; Better tolerability; Paediatrics; Adolescents; Therapeutic drug monitoring; Pharmacokinetics; Cystic Fibrosis; Aspergillosis
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis; Reinfection | interventions — posaconazole; Suspensions

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, multi-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posaconazole arm (Experimental): 90 patients (out of the 135 total patients, therefore with a 2:1 randomization ratio) will receive posaconazole for 12 weeks. Patients in the posaconazole arm will be stratified for body weight and positive sputum cultures for Aspergillus species.
  Patients will be followed-up for a total of 12 months post-randomization.
  Interventions: Drug: Posaconazole 100 MG [Noxafil]; Drug: Posaconazole 40 MG/ML
- Control arm (No Intervention): 45 patients (out of the 135 total patients, therefore with a 2:1 randomization ratio) will not receive the active treatment.
  Patients will be followed-up for a total of 12 months post-randomization. If participants in the control arm are deteriorating during the first 3 months after randomization, it is up to the treating physician to consider treatment for the initial asymptomatic Aspergillus infection

INTERVENTIONS:
Drug: Posaconazole 100 MG [Noxafil] — Posaconazole is a lipophilic, highly permeable triazole, which is practically insoluble in water. Posaconazole inhibits the enzyme CYP51a (also known as Erg11p or lanosterol demethylase). This enzyme is required for catalysation of an essential step in biosynthesis of ergosterol in filamentous fungi and yeasts.
  Posaconazole is favoured over itraconazole and voriconazole with respect to palatability, tolerability and toxicity profile
  Other Names: gastro-resistant tablets Noxafil® 100 mg
  Arms: Posaconazole arm
Drug: Posaconazole 40 MG/ML — Posaconazole is a lipophilic, highly permeable triazole, which is practically insoluble in water. Posaconazole inhibits the enzyme CYP51a (also known as Erg11p or lanosterol demethylase). This enzyme is required for catalysation of an essential step in biosynthesis of ergosterol in filamentous fungi and yeasts.
  Posaconazole is favoured over itraconazole and voriconazole with respect to palatability, tolerability and toxicity profile
  Other Names: 105 ml Noxafil® 40 mg/ml oral suspension
  Arms: Posaconazole arm

SUMMARY:
This study will provide: (1) new insights in the prevalence of Aspergillus infection in children and adolescents with CF aged 8-17 yrs; (2) an in silico modelled dose of posaconazole for children and adolescents with CF and Aspergillus infection aged 8-17 yrs; (3) an intensive sampling PK study to define the optimal dose in a limited number of children and adolescents with CF and Aspergillus infection aged 8-17 yrs; (4) a prospective clinical validation to reduce the residual variability and to allow investigation into PK-PD; and (5) an efficacy evaluation of this dosing regimen to treat Aspergillus infection in children and adolescents with CF to inform future primary efficacy trials.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common inherited life-limiting disease in North European people affecting 90,000 people worldwide with about 45,000 registered in the Patient Registry of the European Cystic Fibrosis Society (ECFS). Progressive lung damage caused by recurrent infection and persistent inflammation is the major determinant of survival with a median age of death at 29 years. Approximately 60% of CF patients are infected with A. fumigatus, a ubiquitous environmental fungus,and its presence is associated with accelerated lung function decline. Half of the patients infected with Aspergillus are <18 years of age. Evidence to guide clinical management of CF-related Aspergillus disease is lacking. A recent survey showed considerable variability in clinical practice among CF consultants. Two-thirds would treat Aspergillus colonization in patients with CF and two-thirds would use an azole antifungal in addition to steroids in the first line treatment of CF-related allergic bronchopulmonary aspergillosis (ABPA). The results of this survey underscore the limited evidence available to guide management of Aspergillus infection in CF.

Posaconazole, being one of the 4 licensed triazole antifungals with good efficacy against Aspergillus species has been chosen as the study drug as it has a better tolerability compared to itraconazole, less toxicity and drug-drug interactions compared to voriconazole and can be administered once daily. Posaconazole is licensed in Europe for the prevention of invasive aspergillus in adult neutropenic patient populations and as salvage therapy for invasive aspergillosis. Several studies have reported on the safety and tolerability of the use of posaconazole in children and adolescents with either haematological malignancies, or chronic granulomatous disease, or those undergoing haematopoietic stem cell transplantation. Currently, no dosing algorithm is available to guide posaconazole dosing in children.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with cystic fibrosis (genetic diagnosis and/or abnormal sweat test and clinical phenotype of lung disease)
2. Age ≥ 8 yrs and < 18 yrs
3. Body weight ≥20 kg
4. Presence of Aspergillus infection as defined for this study
5. Clinically stable condition without a significant change in lung function (FEV1 +/- 10%) or significant worsening of respiratory symptoms over the previous month
6. Able to perform lung function test (FEV1%)
7. Able to produce a sputum sample (spontaneous or induced sputum)
8. Informed Consent given
9. If female and of childbearing age must be using highly effective contraception (and must agree to continue for 7 days after the last dose of investigational medicinal product [IMP]

Exclusion Criteria:

1. Non-CF lung disorder
2. Age < 8 yrs or ≥ 18 yrs
3. Body weight < 20 kg
4. Not able to perform lung function test (FEV1%)
5. Unable to produce a sputum sample (spontaneous or induced sputum)
6. Clinically unstable condition with significant change in lung function or significant worsening of respiratory symptoms
7. Unable to tolerate oral medication
8. Known hypersensitivity to itraconazole or posaconazole, or it's excipients.
9. On active transplant list or transplant recipient
10. Azole resistant Aspergillus sp. cultured
11. Patients receiving terfenadine, ergot alkaloids, astemizole, cisapride, pimozide, halofantrine, quinidine, or HMG-CoA reductase inhibitors metabolised through CYP3A4 (eg. simvastatin, lovastatin, and atorvastatin)
12. Patients receiving omalizumab
13. Received systemic mould-active antifungals in the last month
14. Shortened or elongated QT interval
15. Cardiac failure
16. ALT ≥ 200 U/L
17. AST ≥ 225 U/L
18. Alkaline phosphatase ≥ 460 U/L
19. Bilirubin ≥ 50 umol/L
20. eGFR < 20 ml/min/1.73 m2 (calculated with the Schwartz formula)
21. Patients with known glucose-galactose malabsorption problems
22. Pregnancy2 or breastfeeding
23. Females of childbearing age who do not intend to use contraception measures.
24. Informed Consent not given

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis: Cmax
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis: Cmin
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis:
  Tmax
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis: Area Under the Curve during 1 dosing interval and over 24 hours
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis: Clearance
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis: Distribution volume
Pharmacokinetic parameters of posaconazole | At steady state, day 5-10 of treatment
  The following pharmacokinetic parameter will be calculated using non-compartmental pharmacokinetic analysis: Half-life
Aspergillus isolation from sputum cultures | 3 months after randomisation
  For evaluating the clinical efficacy of posaconazole, the outcome measure that will be analysed is the number of children with negative sputum sample for Aspergillus 3 months after randomisation.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Cmax
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Cmin
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Tmax
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Area Under the Curve
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Clearance
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Distribution volume
Pharmacokinetic parameters of posaconazole | Day 21-35 and day 84 of treatment
  The following pharmacokinetic parameters will be calculated using non-compartmental pharmacokinetic analysis: Half-life
Patients with a favourable clinical response and no signs of Aspergillus infection | 3, 6 and 12 months after randomisation
  Percentage of patients who have a favourable clinical response (defined by pulmonary exacerbation rate, days on antibiotics and corticosteroids, hospital admissions, change in FEV1, change in BMI, CT-chest abnormalities, QoL)
Patients with no signs of Aspergillus infection | 3, 6 and 12 months after randomisation
  Percentage of patients who have no signs of Aspergillus infection (defined by negative sputum cultures and negative serology).
The proportion of participants experiencing AEs and SAEs | Up to 1 year after randomisation
  Assessed according to the Division of AIDS (DAIDS), Table for Grading of the NIAID, NIH, and the US Department of Health and Human Services.

CONTACTS AND LOCATIONS:
Overall Officials: Adilia Warris, Prof, Study Director — University of Exeter
Locations (31):
- Motol University Hospital, Prague, Czechia
- France (3):
  - Centre hospitalier universitaire Dijon Bourgogne, Bourgogne
  - Centre hospitalier universitaire Grenoble Alpes, Grenoble
  - Centre hospitalier universitaire de Montpellier, Montpellier
- Germany (5):
  - Katholisches Klinikum Bochum gGMBH, Klinik für Kinder- und Jugendmedizin der Ruhr-Universität Bochum, St. Josef Hospital, Bochum
  - Technische Universität Dresden, Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Kinder- und Jugendmedizin, Dresden
  - Universitätsklinikum Essen,Pediatric Pulmonology and Cystic Fibrosis Center, Essen
  - Medizinische Hochschule Hannover, Klinik für Pädiatrische Pneumologie, Allergologie und Neonatologie, Hanover
  - Universitätsklinikum Jena, Klinik für Kinder- und Jugendmedizin, Pädiatrische Pneumologie/Allergologie/Mukoviszidose-Zentrum, Jena
- Greece (2):
  - Cystic Fibrosis Department, "Agia Sofia" Children's Hospital, Athens
  - Cystic Fibrosis Center, 3rd Paediatric Dept, Aristotle University of Thessaloniki, Thessaloniki
- Cork University Hospital, Cork, Ireland
- Italy (4):
  - ASST Spedali Civili Paediatric department, Brescia
  - IRCCS Istituto Giannina Gaslini, Genoa
  - University of Parma Department of Medicine and Surgery, Parma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
- Netherlands (4):
  - University Medical Center Groningen (UMCG), Groningen
  - Radboud University Medical Center (RUMC), Nijmegen
  - Erasmus Medical Center (EMC), Rotterdam
  - University Medical Center Utrecht (UMCU), Utrecht
- Centro Hospitalar Universitário Lisboa Norte EPE, Lisbon, Portugal
- Spain (4):
  - Hospital Universitario Materno Infantil Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre,Unidad Multidisciplinar Fibrosis Quística, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- University Children's Hospital Zurich, Zurich, Switzerland
- United Kingdom (5):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University Hospital Nottingham (Queens Medical Centre), Nottingham
  - Sheffield Childrens NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS FT, Southampton
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after the availability of the CSR and therefore from April 2024

REFERENCES:
- [Background] Armstead J, Morris J, Denning DW. Multi-country estimate of different manifestations of aspergillosis in cystic fibrosis. PLoS One. 2014 Jun 10;9(6):e98502. doi: 10.1371/journal.pone.0098502. eCollection 2014. PMID 24914809
- [Background] Rowbotham NJ, Smith S, Prayle AP, Robinson KA, Smyth AR. Gaps in the evidence for treatment decisions in cystic fibrosis: a systematic review. Thorax. 2019 Mar;74(3):229-236. doi: 10.1136/thoraxjnl-2017-210858. Epub 2018 Oct 9. PMID 30301819
- [Background] Boyle M, Moore JE, Whitehouse JL, Bilton D, Downey DG. The diagnosis and management of respiratory tract fungal infection in cystic fibrosis: A UK survey of current practice. Med Mycol. 2019 Feb 1;57(2):155-160. doi: 10.1093/mmy/myy014. PMID 29554296
- [Background] Welzen ME, Bruggemann RJ, Van Den Berg JM, Voogt HW, Gilissen JH, Pajkrt D, Klein N, Burger DM, Warris A. A twice daily posaconazole dosing algorithm for children with chronic granulomatous disease. Pediatr Infect Dis J. 2011 Sep;30(9):794-7. doi: 10.1097/INF.0b013e3182195808. PMID 21772229
- [Background] Groll AH, Abdel-Azim H, Lehrnbecher T, Steinbach WJ, Paschke A, Mangin E, Winchell GA, Waskin H, Bruno CJ. Pharmacokinetics and safety of posaconazole intravenous solution and powder for oral suspension in children with neutropenia: an open-label, sequential dose-escalation trial. Int J Antimicrob Agents. 2020 Sep;56(3):106084. doi: 10.1016/j.ijantimicag.2020.106084. Epub 2020 Jul 17. PMID 32682946
- [Background] King J, Brunel SF, Warris A. Aspergillus infections in cystic fibrosis. J Infect. 2016 Jul 5;72 Suppl:S50-5. doi: 10.1016/j.jinf.2016.04.022. Epub 2016 May 11. PMID 27177733
- [Background] Periselneris J, Nwankwo L, Schelenz S, Shah A, Armstrong-James D. Posaconazole for the treatment of allergic bronchopulmonary aspergillosis in patients with cystic fibrosis. J Antimicrob Chemother. 2019 Jun 1;74(6):1701-1703. doi: 10.1093/jac/dkz075. PMID 30805605
- [Background] Dolton MJ, Bruggemann RJ, Burger DM, McLachlan AJ. Understanding variability in posaconazole exposure using an integrated population pharmacokinetic analysis. Antimicrob Agents Chemother. 2014 Nov;58(11):6879-85. doi: 10.1128/AAC.03777-14. Epub 2014 Sep 8. PMID 25199779
- [Background] Castellani C, Duff AJA, Bell SC, Heijerman HGM, Munck A, Ratjen F, Sermet-Gaudelus I, Southern KW, Barben J, Flume PA, Hodkova P, Kashirskaya N, Kirszenbaum MN, Madge S, Oxley H, Plant B, Schwarzenberg SJ, Smyth AR, Taccetti G, Wagner TOF, Wolfe SP, Drevinek P. ECFS best practice guidelines: the 2018 revision. J Cyst Fibros. 2018 Mar;17(2):153-178. doi: 10.1016/j.jcf.2018.02.006. Epub 2018 Mar 3. PMID 29506920
- [Background] Patel D, Popple S, Claydon A, Modha DE, Gaillard EA. Posaconazole therapy in children with cystic fibrosis and Aspergillus-related lung disease. Med Mycol. 2020 Jan 1;58(1):11-21. doi: 10.1093/mmy/myz015. PMID 30877757
- [Background] Krishna G, Ma L, Martinho M, Preston RA, O'Mara E. A new solid oral tablet formulation of posaconazole: a randomized clinical trial to investigate rising single- and multiple-dose pharmacokinetics and safety in healthy volunteers. J Antimicrob Chemother. 2012 Nov;67(11):2725-30. doi: 10.1093/jac/dks268. Epub 2012 Jul 24. PMID 22833639
- [Background] Tragiannidis A, Herbruggen H, Ahlmann M, Vasileiou E, Gastine S, Thorer H, Frohlich B, Muller C, Groll AH. Plasma exposures following posaconazole delayed-release tablets in immunocompromised children and adolescents. J Antimicrob Chemother. 2019 Dec 1;74(12):3573-3578. doi: 10.1093/jac/dkz359. PMID 31504563